CLINICAL TRIAL: NCT00684294
Title: Phase I Trial of TGFB2-Antisense-GMCSF Gene Modified Autologous Tumor Cell (TAG) Vaccine for Advanced Cancer
Acronym: Auto TAG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Since no safety issues have been reported to date in association with TAG vaccine, no further survival follow-up will be done.
Sponsor: Mary Crowley Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCMRC #08-08
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Advanced Metastatic
Keywords: cancer; oncology; solid tumor
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — Product Labeling; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAG Vaccine 1 x 10^7 cells/ injection (Experimental): TAG Vaccine 1 x 10^7 cells/injection
  Interventions: Biological: TGFβ2 Antisense-GMCSF Gene Modified Autologous Tumor Cell (TAG) Vaccine
- TAG Vaccine 2.5 X 10^7 cells/injection (Experimental): TAG Vaccine 2.5 X 10^7 cells/injection
  Interventions: Biological: TGFβ2 Antisense-GMCSF Gene Modified Autologous Tumor Cell (TAG) Vaccine

INTERVENTIONS:
Biological: TGFβ2 Antisense-GMCSF Gene Modified Autologous Tumor Cell (TAG) Vaccine — Patients with solid tumors will receive TAG Vaccine 1 x 10^7 cells/ injection or TAG Vaccine 2.5 X 10^7 cells/injection once a month for up to 12 doses via intradermal injection as long as sufficient material is available. Selection of cohort is dependent on the amount of tumor cell yield following harvest and processing.

SUMMARY:
Preliminary studies with a variety of vaccines suggest target accessibility (potential immunogenicity) in a variety of solid tumors to immune directed approaches. However, four primary factors limit the generation of effective immune mediated anticancer activity in therapeutic application:

1. identifying and/or targeting cancer associated immunogen(s) in an individual patient
2. insufficient or inhibited level of antigen presenting cell priming and/or presentation
3. suboptimal T cell activation and proliferation
4. cancer-induced inhibition of the anticancer immune response in both afferent and efferent limbs.

In an effort to overcome these limitations, we have designed a novel autologous vaccine to address inability to fully identify cancer associated antigens, antigen recognition by the immune system (i.e. antigen to immunogen), effector potency, and cancer-induced resistance. We have completed clinical investigations using two different gene vaccine approaches to induce enhancement of tumor antigen recognition which have demonstrated therapeutic efficacy. Specifically, both the use of a GMCSF gene transduced vaccine and a TGFβ2 antisense gene vaccine, in separate trials, have demonstrated similar beneficial effects without any evidence of significant toxicity in advanced cancer patients. The GMCSF transgene directly stimulates increased expression of tumor antigen(s) and enhances dendritic cell migration to the vaccination site. TGFβ2 blockade following intracellular TGFβ2 antisense gene expression reduces production of immune inhibiting activity at the vaccine site. These agents have never been used in combination but the rationale of integrating enhancement of an anticancer immune response concurrently with a reduction in cancer-induced immune suppression is conceptually sound. We will harvest autologous cancer cells from patients with advanced refractory cancer. We have constructed a TGFβ2 antisense / GMCSF expression vector plasmid and have successfully demonstrated preclinical activity of the vector function following transfection by electroporation and irradiation of autologous cancer tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic non-curable solid tumor (if limited to a single lesion and not a candidate for curative surgery or radiation therapy).
* Completed ≥1 conventional therapy.
* Clinically indicated surgery or procedure to collect available tumor in sufficient quantity ("golf ball size," pleural or ascites fluid may also be collected) for vaccine processing.
* Subjects that have completed all acceptable therapies that are the current standard of care for their respective diseases.
* Recovered from all toxicities related to prior therapies.
* Subjects with brain metastases treated at least ≥2 months prior to enrollment, without related clinical symptoms and must have a stable neurological exam on the screening evaluation.
* ≥1 measurable or evaluable lesion.
* Age ≥18 years.
* ECOG performance status (PS) 0-1.
* Normal organ and marrow function:

  * Absolute granulocyte count: ≥1,500/mm3
  * Platelets: ≥100,000/mm3
  * Total bilirubin: ≤2 mg/dL
  * AST(SGOT)/ALT(SGPT): ≤2x institutional upper limit of normal
  * Creatinine: <1.5 mg/dL
* Ability to understand and the willingness to sign a written informed consent document.
* Negative pregnancy test.

Exclusion Criteria:

* Surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to entering the study.
* Patient must not have received any other investigational agents within 30 days prior to study entry.
* Patients with known brain metastases unless treated and stable for ≥2 months.
* Patients with mucinous adenocarcinoma.
* Short term (<30 days) concurrent systemic steroids ≤ 0.125 mg/kg prednisone per day (maximum 10 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded. Patients requiring steroids following previous CNS radiation for metastatic disease are excluded.
* Prior splenectomy.
* Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for ≥2 years.
* Kaposi's Sarcoma.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or nursing.
* Patients who are HIV positive.
* Patients with chronic Hepatitis B and C infection.
* Patients with a history of autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-05-27 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
To determine safety following the administration of TAG vaccine in advanced solid tumor patients who have no acceptable form of standard therapy. | 6 months

SECONDARY OUTCOMES:
To determine the time to progression following the administration of TAG vaccine. | survival
To evaluate the effect on immune stimulation. | baseline, Month 3, and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States